CLINICAL TRIAL: NCT04149795
Title: Physical Activity Recommendation Behaviour in German Psychologists
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Moritz Petzold, Principal Investigator, Charite University, Berlin, Germany
Other Study IDs: PAR_P
Record Dates: First submitted 2019-10-30; First posted 2019-11-04 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Mental Disorder; Physical Activity
Keywords: Physical activity; Mental disorder; Recommendation behaviour; Prescription Behaviour; Mental health; Exercise
MeSH Terms: conditions — Mental Disorders; Motor Activity; Psychological Well-Being

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Clinical psychologists in Germany: Clinical psychologists in Germany currently working with patients with mental disorders
  Interventions: Diagnostic Test: Online questionnaire

INTERVENTIONS:
Diagnostic Test: Online questionnaire — Online questionnaire via SoSciSurvey

SUMMARY:
The purpose of this study is to examine the physical activity recommendation behaviour, beliefs, barriers and exercise participation in German psychologists working with patients with mental disorders.

DETAILED DESCRIPTION:
Physical activity plays an important role in the prevention and treatment of mental disorders. Despite the potential mental health benefits, large proportions of patients with mental disorders do not meet the physical activity recommendations.

Clinical psychologists play a key role in the recommendation of physical activity to their patients. There are no previous studies that examine physical activity recommendation behaviour in German psychologists.

The purpose of this study is to examine the physical activity recommendation behaviour, beliefs, barriers and exercise participation in German psychologists working with patients with mental disorders.

ELIGIBILITY:
Inclusion Criteria:

* Clinical psychologist
* Currently working with patients with mental disorders
* At least 18 years old
* Sufficient German skills for answering the questionnaire

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Clinical psychologists that currently work with patients with mental disorders in Germany.
Sampling Method: Non-Probability Sample
Enrollment: 454 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2020-04-25 (Actual); Study Completion 2020-04-25 (Actual)

PRIMARY OUTCOMES:
Exercise in Mental Illness Questionnaire (EMIQ) - German Version | 1 day
  Questionnaire assessing the following areas: knowledge, beliefs, behaviours regarding and participation in physical activity in mental health professionals.

CONTACTS AND LOCATIONS:
Overall Officials: Moritz B Petzold, Dipl.-Psych., Principal Investigator — Charité Universitätsmedizin Berlin- Charité Campus Mitte - Department for Psychiatry and Psychotherapy
Locations (1):
- Charité Universitätsmedizin Berlin - Department for Psychiatry and Psychotherapy - Charité Campus Mitte, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided